CLINICAL TRIAL: NCT01892696
Title: Arterial Pulse Pressure Variation and Inferior Vena Cava Distensibility Affected by Inspiratory Flow Waveforms in Mechanically Ventilated Patients: Time for a Change
Brief Title: Effects of Inspiratory Flow Waveforms on Preload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Principal Investigator, Hajjej Zied, Dr, Military Hospital of Tunis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CvDVPPIVC; CvD1977 (Other: Military Hospital of Tunis)
Record Dates: First submitted 2013-06-26; First posted 2013-07-04 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Cardiac Output, Low
Keywords: inspiratory flow pattern; mechanical ventilation; cardiac preload; arterial pulse pressure variation; inferior vena cava collapsibility
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mechanically ventilated patients (Other): patients admitted to a 18-bed medical surgical intensive care unit of the military hospital of Tunisia and were mechanically ventilated fully adapted to their ventilator and in sinus rhythm.
  intervention:varying inspiratory flow waveforms
  Interventions: Device: varying inspiratory flow waveforms

INTERVENTIONS:
Device: varying inspiratory flow waveforms — inspiratory flow waveform was changed, in a randomized sequence using a computer ,to one of the following modalities: 1) constant inspiratory flow; 2) decelerating inspiratory flow Each inspiratory flow waveform was maintained for 30 min. During the last 5 min of this period the physiological signals were collected and measures were performed.

SUMMARY:
The clinical usefulness of inspiratory flow pattern manipulation during mechanical ventilation remains unclear. The aim of this study was to investigate the effects of different inspiratory flow waveforms, i.e. constant and decelerating, on cardiac preload in mechanically ventilated patients assessed by arterial pulse pressure variation (PPV) and inferior vena cava distensibility.

DETAILED DESCRIPTION:
During mechanical ventilation the lungs can be inflated with different pressure and flow waveforms. Originally the piston-driven mechanical ventilators generated a quasi-sinusoidal flow waveform, whereas the newer electronically controlled ventilators can also produce constant and decelerating waveforms. According to several theoretical,animal and clinical studies,the inspiratory flow waveform affects the distribution of the inspired gas as well as respiratory mechanics and gas exchange. However, other studies failed to show any significant effect.But there is no study interested to the effects of inspiratory flow waveforms on cardiac preload. Thus, the clinical usefulness of inspiratory flow pattern manipulation remains unclear, though the capacity for selection of different inspiratory flow waveforms is provided by most modern, microprocessor-equipped ventilators. Therefore, the purpose of this study was to compare the effects of flow patterns (sinusoidal, constant and decelerating) on dynamic measurements of cardiac preload dependence such as arterial pulse pressure variation (ΔPP) and distensibility index of the inferior vena cava (dIVC).

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation
* Volume AssistControl Ventilation
* sinus rhythm

Exclusion Criteria:

* pressure mode
* arrhythmia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
change in pulse pressure variation (ΔPP) and distensibility index of the inferior vena cava (dIVC)when varying inspiratory flow waveforms | 2h
  Each inspiratory flow waveform was maintained for 30 min with 60 minutes washout period

CONTACTS AND LOCATIONS:
Overall Officials: zied hajjej, Dr, Principal Investigator — Military Hospital of Tunis
Locations (1):
- Military hospital of tunis, Tunis, Mont Fleury, Tunisia